CLINICAL TRIAL: NCT00993551
Title: Timing of Primary Surgery for Cleft Palate
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Munro (Other)
Collaborators: University of Liverpool (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Copenhagen (Other); Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Kevin Munro, Professor of Audiology, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-017-E; 1U01DE018837-01A1 (NIH); Sponsor Reference: 57201 (Other: The University of Manchester (UK)); NIHR Portfolio Reference 30200 (Other: NIHR)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Cleft Palate
Keywords: cleft palate; paediatric; pediatric; surgery; speech; velopharyngeal
MeSH Terms: conditions — Cleft Palate; Speech | interventions — cyclopropapyrroloindole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 month surgery (Experimental): Infants will receive primary surgery at age 12 months using Sommerlad technique
  Interventions: Procedure: primary surgery for cleft palate
- 6 month surgery (Experimental): Infants will receive primary surgery at age 6 months using Sommerlad technique.
  Interventions: Procedure: primary surgery for cleft palate

INTERVENTIONS:
Procedure: primary surgery for cleft palate — Surgery completed using the Sommerlad technique

SUMMARY:
This trial is a randomised controlled trial with a parallel design taking place in centres across the UK, Scandinavia and Brazil.

650 infants with a diagnosis of isolated cleft palate who are considered medically fit for operation at 6 months, and who meet the inclusion criteria, will be included in the trial and randomised to receive either:

* Surgery at age 6 months, OR
* Surgery at age 12 months.

The main objective is to determine whether surgery for cleft palate, using a Sommerlad technique, at age 6 months, when compared to surgery using the same technique at age 12 months, improves velopharyngeal function at age 5 years. All infants will be followed up at age 12 months, 3 years and five years for the assessment of the primary outcomes( at age 5 years) and secondary outcomes.

DETAILED DESCRIPTION:
Infants will be followed up at age 12 months, 3 years and five years. At each visit the following will be assessed:

Age 12 months

* Speech development (canonical babbling)
* Audiological assessments
* Growth

Age 3 years

* Speech development
* Audiological assessments

Age 5 Years

* Speech development
* Audiological assessments
* Dentofacial development (Soft Tissue ANB and Maxillary arch constriction score using modified Huddart Bodenham scoring)

ELIGIBILITY:
Inclusion Criteria:

* Infants with isolated cleft palate
* Medically fit for operation at 6 months, corrected for gestational age
* Written informed proxy consent
* One parent/carer a native language speaker in the country of residence

Exclusion Criteria:

* Consent not obtained
* b. Infants with syndromic cleft palate (except Van der Woude syndrome, which can be included if hearing is not affected) or severe developmental delay
* Congenital sensorineural hearing loss or middle ear anomalies;
* Variation in the anatomical presentation is such that the surgeon who will perform the procedure considers that one stage closure with the Sommerlad technique would be inappropriate;
* Submucous cleft palate (defined by the classical triad of signs, bifid, uvula, bony defect of the hard palate, muscular diastasis, as described by Jensen et al (1988).
* Where the language spoken at home is not the majority language in the country of residence.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 558 (Actual)
Dates: Start 2010-07; Primary Completion 2020-08 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for the TOPS trial is insufficient velopharyngeal function. | 5 years
  Unit of measure: Sufficient (VPC sum <=3) or insufficient (VPC sum>=4). VPC sum measured on scale from 1 to 6.

SECONDARY OUTCOMES:
Velopharyngeal function;1.Velopharyngeal composite score summary (VPC sum) 2.Insufficient velopharyngeal function (VPC rate) | 3 and 5 years
  Velopharyngeal function measured by combination of VPC sum and VPC rate. VPC sum is measured as for primary outcome measure and VPC rate on a 3 point scale; insufficient, marginal or sufficient
Velopharyngeal function: Velopharyngeal insufficiency symptoms | 3 years
  It will be measured either by presence of resonance "yes" within normal limit or "no" if not within normal limit
Canonical babbling; 1.Canonical babbling present 2.Canonical babbling ratio | 12 months
  Canonical babbling is measured by presence of vocalised syllables and percentage ( ratio) of children vocalising canonical or non canonical babbling of syllables
Canonical babbling; 3.Consonant inventory | 12 months
  Consonant inventory is measured by the number of correct sounds produced
Articulation: 1. Percent consonant correct (PCC) | 3 and 5 years
  Articulation is measured by the percentage of children vocalising the correct consonants
Articulation: 1.Percent Correct Placement (PCP) 3. Percent Correct Manner (PCM) 4. Non-oral consonant errors 5. Oral consonant errors | 3 and 5 years
  Articulation is measured by the percentage of children vocalising correct consonants ( oral and non-oral) in the correct placement and manner
Postoperative/long term complications | 48 hours and 30 days postoperatively
  Complications are measured by assessment for presence (yes or no) of the following:1.Dehiscence 2.Infection 3.Evidence of fistula
Postoperative/long term complications | at 3 and 5 year follow up
  measured by assessment for presence (yes or no) or evidence of fistula
Hearing: hearing level assessment | 12 months
  Assessment of hearing level by Tympanometry and abnormal transient otoacoustic emission (TEOAE)
Hearing level assessment for: 1. Abnormal Puretone audiometry in one and or both ears. | 3 and 5 years
  Hearing level is assessed by Puretone audiometry
Hearing level assessment | 3 and 5 years
  Severity of hearing loss is measured in better ear is categorised as normal, mild, moderate, severe or profound.
Middle ear function | 12 months, 3 and 5 years
  Middle ear function is assessed by presence of flat line Tympanogram in at least one ear and or both ears
Dentofacial development: Soft tissue ANB (the angle between soft tissue nasion, | 5 years
  Soft tissue development is measured by measuring the angle between two points (SSs-ns-sms) on a profile photograph. The unit of measure is angular degrees
Dentofacial development; Maxillary arch constriction score | 5 years
  This outcome is assesed using modified Huddart/Bodenham scoring system which is a range from -24 to +8
Growth assessment for nude weight | 12 months
  Growth is measured in Kg body weight in nude
Growth Assessment for crown to heel length and occipitofrontal circumference | 12 months
  Assessment for crown to heel length and Occipitofrontal circumference are in centimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Munro, Principal Investigator — University of Manchester
Locations (23):
- University of Sao Paulo, Bauru, Brazil
- Denmark (2):
  - Århus Speech and Hearing Institute, Aarhus
  - Copenhagen Cleft Palate Centre, Copenhagen
- Norway (2):
  - Helse Bergen HF, Bergen
  - Oslo University Hospital, Oslo
- Sweden (6):
  - Göteborg University, Gothenburg
  - University of Linköping, Linköping
  - Malmö University Hospital, Malmo
  - Karolinska University Hospital, Stockholm
  - Umeå University, Umeå
  - Uppsala University, Uppsala
- United Kingdom (12):
  - Belfast Health and Social Care Trust, Belfast
  - Birmingham Children's NHS Foundation Trust, Birmingham
  - North Bristol NHS Foundation Trust, Bristol
  - Edinburgh Hospital for Sick Children, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - Leeds University Hospitals NHS foundation Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Manchester University NHS Foundation Trust, Manchester
  - Newcastle University Hospitals NHs Foundation Trust, Newcastle
  - Oxford University Hospitals NHS Trust, Oxford
  - Salisbury District Hospital, Salisbury
  - Abertawe Bro Morgannwg University Health Board, Swansea

REFERENCES:
- [Derived] Gamble C, Persson C, Willadsen E, Albery L, Soegaard Andersen H, Zattoni Antoneli M, Appelqvist M, Aukner R, Bodling P, Bowden M, Brunnegard K, Cairns G, Calladine S, Campbell L, Clayton-Smith J, Cooper R, Conroy E, El-Angbawi A, Kildegaard Emborg B, Enfalt Wikman J, Fitzpatrick B, Fukushiro AP, Guedes de Azevedo Bento Goncalves C, Havstam C, Hvistendahl AK, Jorgensen LD, Klinto K, Berntsen Kvinnsland M, Larham C, Lemvik J, Leturgie L, Liljerehn E, Lodge N, Lohmander A, McMahon S, Mehendale F, Miguel HC, Moe M, Nielsen JB, Nyberg J, Pedersen NH, Phippen G, Alvarez Piazentin-Penna SH, Patrick K, Pliskin L, Rigby L, Semb G, Southby L, Sporre M, Bjorkman Taleman AS, Tangstad J, Trindade IEK, Underwood I, van Eeden S, Westberg LR, Williamson PR, Paciello Yamashita R, Munro K, Walsh T, Shaw W; TOPS Study Group. Timing of Primary Surgery for Cleft Palate. N Engl J Med. 2023 Aug 31;389(9):795-807. doi: 10.1056/NEJMoa2215162. PMID 37646677
- [Derived] Willadsen E, Cooper R, Conroy E, Gamble C, Albery L, Andersen H, Appelqvist M, Bodling P, Bowden M, Brunnegard K, Enfalt J, van Eeden S, Goncalves C, Fukushiro A, Jorgensen L, Lemvik J, Leturgie L, Liljerehn E, Lodge N, McMahon S, Miguel H, Patrick K, Phippen G, Piazentin-Penna S, Southby L, Taleman AS, Tangstad J, Yamashita R, Shaw W, Munro K, Walsh T, Persson C. Inter-rater reliability in classification of canonical babbling status based on canonical babbling ratio in infants with isolated cleft palate randomised to Timing of Primary Surgery for Cleft Palate (TOPS). Clin Linguist Phon. 2023 Jan 2;37(1):77-98. doi: 10.1080/02699206.2021.2012259. Epub 2022 Jan 31. PMID 35100923
- [Derived] Conroy EJ, Cooper R, Shaw W, Persson C, Willadsen E, Munro KJ, Williamson PR, Semb G, Walsh T, Gamble C; TOPS trial management group. A randomised controlled trial comparing palate surgery at 6 months versus 12 months of age (the TOPS trial): a statistical analysis plan. Trials. 2021 Jan 4;22(1):5. doi: 10.1186/s13063-020-04886-y. PMID 33397459
- [Derived] Shaw W, Semb G, Lohmander A, Persson C, Willadsen E, Clayton-Smith J, Trindade IK, Munro KJ, Gamble C, Harman N, Conroy EJ, Weichart D, Williamson P. Timing Of Primary Surgery for cleft palate (TOPS): protocol for a randomised trial of palate surgery at 6 months versus 12 months of age. BMJ Open. 2019 Jul 11;9(7):e029780. doi: 10.1136/bmjopen-2019-029780. PMID 31300507